CLINICAL TRIAL: NCT02078973
Title: The Effects of Tolvaptan on Renal Handling of Water and Sodium, Vasoactive Hormones and Circulatory System, During Basal Conditions and During Inhibition of the Nitric Oxide System in Healthy Subjects. A Dose-response Study.
Brief Title: Effect of the Aquaretic Tolvaptan on Nitric Oxide System. A Dose-response Study (DOVA)
Acronym: DOVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, Professor, MD, Dr.Sci., Regional Hospital Holstebro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SAFA-1-2014; 2013-003800-38 (EudraCT Number)
Record Dates: First submitted 2014-03-01; First posted 2014-03-05 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Nephropathy
Keywords: Tolvaptan; L-NMMA; Healthy subjects; Nephrology
MeSH Terms: conditions — Kidney Diseases | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 15 mg tolvaptan (Active Comparator): Oral administration of 15 mg tolvaptan on each examination day.
  Interventions: Drug: 15 mg tolvaptan
- 30 mg tolvaptan (Active Comparator): Oral administration of 30 mg tolvaptan on each examination day.
  Interventions: Drug: 30 mg tolvaptan
- 45 mg tolvaptan (Active Comparator): Oral administration of 45 mg tolvaptan on each examination day.
  Interventions: Drug: 45 mg tolvaptan
- Placebo (Placebo Comparator): Oral administration of a Unikalk tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 15 mg tolvaptan — 15 mg pr day for 1 day
  Other Names: Samsca
  Arms: 15 mg tolvaptan
Drug: 30 mg tolvaptan — 30 mg pr day for 1 day
  Other Names: Samsca
  Arms: 30 mg tolvaptan
Drug: 45 mg tolvaptan — 45 mg pr day for 1 day
  Other Names: Samsca
  Arms: 45 mg tolvaptan
Drug: Placebo — 1 tablet Unikalk pr day for 1 day
  Other Names: Unikalk
  Arms: Placebo

SUMMARY:
Tolvaptan is a selective vasopressin receptor antagonist (V2R) that increases free water and sodium excretion. Inhibition of V2R increases vasopressin concentration in plasma, which stimulates V1-receptors in the vascular bed and may change both central and brachial hemodynamics and plasma concentration of vasoactive hormones.

The purpose of the study is to measure the effects of tolvaptan on renal handling of water and sodium, systemic hemodynamics and vasoactive hormones at baseline and during nitric oxide (NO)-inhibition with L-NG-monomethyl-arginine (L-NMMA).

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18-40 years
* Body Mass Index (BMI) 18,5-30 kg/m2

Exclusion Criteria:

* Anamnestic or clinical signs of heart, lung, lever, kidney and brain disease
* Neoplastic disease
* Drug abuse
* Alcohol abuse
* Medical treatment except peroral anticontraceptive
* Pregnancy
* Smoking
* Abnormal blood and urine sample
* Abnormal ECG
* Blood donation within a month before examination
* Arterial hypertension (>140 mmHg systolic and/or 90 mmHg diastolic)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
CH2O | 5-6 Hours
  Measurement of H2O clearance at baseline, during and after L-NMMA infusion

SECONDARY OUTCOMES:
Urine biomarkers(Aquaporins and Epithelial Sodium Channels γ) | 5-6 Hours
Central and brachial blood pressure | 5-6 Hours
Augmentation Index | 5-6 Hours
Vasoactive Hormones( Angiotensin II, Aldosterone, Endothelin, Atrial Natriuretic Peptide, Brain Natriuretic Peptide, Arginin Vasopressin) | 5-6 Hours
Fractional sodium excretion | 5-6 Hours
  Measurement of Sodium excretion at baseline, during and after L-NMMA infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Frank H Mose, MD, PhD, Principal Investigator — Department of medical research
Locations (1):
- Department of medical research, Holstebro, Denmark

REFERENCES:
- [Derived] Al Therwani S, Rosenbaek JB, Mose FH, Bech JN, Pedersen EB. Effect of tolvaptan on renal water and sodium excretion and blood pressure during nitric oxide inhibition: a dose-response study in healthy subjects. BMC Nephrol. 2017 Mar 13;18(1):86. doi: 10.1186/s12882-017-0501-1. PMID 28288570